CLINICAL TRIAL: NCT05758909
Title: Evaluation of the Viability and Safety of Early Discharge Protocol After TAVI Implantation
Acronym: FAST TRACK
Status: Active, not recruiting | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: EPIC19-FAST TRACK
Record Dates: First submitted 2023-02-05; First posted 2023-03-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Aortic Valve Disease; Aortic Valve Stenosis; Heart Valve Diseases
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving transfemoral (TF) TAVI: TF TAVI
  Interventions: Device: TF TAVI

INTERVENTIONS:
Device: TF TAVI — Follow-up Observation of patients having received a TF-TAVI

SUMMARY:
Evaluation of the safety and efficacy of early discharge (24 hours) after transfemoral transcatheter aortic prosthesis implantation (TAVI).

DETAILED DESCRIPTION:
Evaluation of the safety and efficacy of early discharge (24 hours) after transfemoral transcatheter aortic prosthesis implantation (TAVI).

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following conditions will be included:

* Patients ≥ 18 years undergoing transfemoral TAVI implantation scheduled, performed on an outpatient basis.
* Patients with percutaneous implant.
* Patients undergoing the procedure under superficial sedation or Local anesthesia.
* Patients with baseline narrow QRS that does not change after implantation, or definitive pacemaker carrier.
* Patients who have signed the informed consent.

Exclusion Criteria:

Patients who do not meet any of the following conditions:

* Patients with a wide QRS (greater than or equal to 120 msec) at baseline, with the except for patients with permanent pacemakers.
* Hospitalized patients undergoing urgent TAVI implantation.
* Patients with access other than percutaneous transfemoral.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing scheduled transfemoral TAVI implantation, performed on an outpatient basis
Sampling Method: Probability Sample
Enrollment: 585 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of early safety | 30 days
  Proportion of patients with early safety defined as:
  * Cardiovascular death.
  * Stroke.
  * Myocardial Infarction.
  * Hospitalization for any reason .
  * Major vascular complications.
  * Need for pacemakers.

SECONDARY OUTCOMES:
Assessment of Cardiovascular death | 30 days
  Assessment of Cardiovascular death
Assessment of Cardiovascular death | 12 months
  Assessment of Cardiovascular death
Assessment of Stroke | 30 days
  Incidence of patients with stroke diagnosed by a Neurologist according to VARC 3 criteria
Assessment of Stroke | 12 months
  Incidence of patients with stroke diagnosed by a Neurologist according to VARC 3 criteria
Assessment of Myocardial Infarction | 30 days
  Incidence of patients with Myocardial Infarction diagnosed by Cardiologist according to VARC 3 criteria
Assessment of Myocardial Infarction | 12 months
  Incidence of patients with Myocardial Infarction diagnosed by Cardiologist according to VARC 3 criteria
Assessment of Hospitalization for any reason | 30 days
  Incidence of patients with Hospitalization for any reason according to VARC 3 criteria
Assessment of Hospitalization for any reason | 12 months
  Incidence of patients with Hospitalization for any reason according to VARC 3 criteria
Assessments of Major Vascular Complications | 30 days
  Incidence of patients with Major Vascular Complications according to VARC 3 criteria
Assessments of Major Vascular Complications | 12 months
  Incidence of patients with Major Vascular Complications according to VARC 3 criteria
Assessments of need for pacemakers | 30 days
  Incidence of patients with need for pacemakers according to VARC 3 criteria
Assessments of need for pacemakers | 12 months
  Incidence of patients with need for pacemakers according to VARC 3 criteria
Assessment of hospitalization time | at discharge
  Incidence of patients with hospitalization according to VARC 3 criteria
Assessment of hospitalization due cardiac reasons | 12 months
  Incidence of patients with hospitalization due cardiac reasons according to VARC 3 criteria
Assessment of hospitalization due cardiac reasons | 30 days
  Incidence of patients with hospitalization due cardiac reasons according to VARC 3 criteria

CONTACTS AND LOCATIONS:
Locations (13):
- Spain (13):
  - Hospital Universitario A Coruña, A Coruña
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Clinico San Carlos, Aravaca
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital de Santa Creu I Sant Pau, Barcelona
  - Hospital Universitari Vall Hebron, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari i Politècnic la Fe, Valencia

REFERENCES:
- [Background] Barbanti M, van Mourik MS, Spence MS, Iacovelli F, Martinelli GL, Muir DF, Saia F, Bortone AS, Densem CG, van der Kley F, Bramlage P, Vis M, Tamburino C. Optimising patient discharge management after transfemoral transcatheter aortic valve implantation: the multicentre European FAST-TAVI trial. EuroIntervention. 2019 Jun 20;15(2):147-154. doi: 10.4244/EIJ-D-18-01197. PMID 30777842
- [Background] van Gils L, Baart S, Kroon H, Rahhab Z, El Faquir N, Rodriguez Olivares R, Aga Y, Maugenest AM, Theuns DA, Boersma E, Szili Torok T, De Jaegere PP, Van Mieghem NM. Conduction dynamics after transcatheter aortic valve implantation and implications for permanent pacemaker implantation and early discharge: the CONDUCT-study. Europace. 2018 Dec 1;20(12):1981-1988. doi: 10.1093/europace/euy074. PMID 29688322
- [Background] Aldalati O, Keshavarzi F, Kaura A, Byrne J, Eskandari M, Deshpande R, Monaghan M, Wendler O, Dworakowski R, MacCarthy P. Factors associated with safe early discharge after transcatheter aortic valve implantation. Cardiol J. 2018;25(1):14-23. doi: 10.5603/CJ.a2017.0087. Epub 2017 Jul 17. PMID 28714522
- [Background] Serletis-Bizios A, Durand E, Cellier G, Tron C, Bauer F, Glinel B, Dacher JN, Cribier A, Eltchaninoff H. A Prospective Analysis of Early Discharge After Transfemoral Transcatheter Aortic Valve Implantation. Am J Cardiol. 2016 Sep 15;118(6):866-872. doi: 10.1016/j.amjcard.2016.06.035. Epub 2016 Jun 27. PMID 27453514
- [Background] Chandrasekhar J, Mehran R. Same or next day discharge: A new chapter in transcatheter aortic valve implantation. Catheter Cardiovasc Interv. 2016 Jan 1;87(1):143-4. doi: 10.1002/ccd.26388. PMID 27410958
- [Background] Wood DA, Lauck SB, Cairns JA, Humphries KH, Cook R, Welsh R, Leipsic J, Genereux P, Moss R, Jue J, Blanke P, Cheung A, Ye J, Dvir D, Umedaly H, Klein R, Rondi K, Poulter R, Stub D, Barbanti M, Fahmy P, Htun N, Murdoch D, Prakash R, Barker M, Nickel K, Thakkar J, Sathananthan J, Tyrell B, Al-Qoofi F, Velianou JL, Natarajan MK, Wijeysundera HC, Radhakrishnan S, Horlick E, Osten M, Buller C, Peterson M, Asgar A, Palisaitis D, Masson JB, Kodali S, Nazif T, Thourani V, Babaliaros VC, Cohen DJ, Park JE, Leon MB, Webb JG. The Vancouver 3M (Multidisciplinary, Multimodality, But Minimalist) Clinical Pathway Facilitates Safe Next-Day Discharge Home at Low-, Medium-, and High-Volume Transfemoral Transcatheter Aortic Valve Replacement Centers: The 3M TAVR Study. JACC Cardiovasc Interv. 2019 Mar 11;12(5):459-469. doi: 10.1016/j.jcin.2018.12.020. PMID 30846085